CLINICAL TRIAL: NCT06202079
Title: A Phase 2 Clinical Trial Comparing the Efficacy and Safety of Once-weekly GZR4 Injection Versus Once-daily Insulin Degludec in Subjects with Type 2 Diabetes Mellitus on OAD Therapy or OAD Therapy in Combination with Basal Insulin
Brief Title: A Trial Comparing the Efficacy and Safety of GZR4 Injection Versus Insulin Degludec in Subjects with Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GL-GZR-CH2007
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GZR4 Injection (Experimental): GZR4 Injection + Oral Antidiabetic Drug
  Interventions: Drug: GZR4 Injection
- Insulin Degludec (Active Comparator): Insulin Degludec + Oral Antidiabetic Drug
  Interventions: Drug: Insulin Degludec

INTERVENTIONS:
Drug: GZR4 Injection — GZR4 injection s.c., once-weekly, treat-to-target dose
  Arms: GZR4 Injection
Drug: Insulin Degludec — Insulin Degludec s.c., once-daily, treat-to-target dose
  Arms: Insulin Degludec

SUMMARY:
This study compares the efficacy, safety, and tolerability of once-weekly GZR4 Injection versus once-daily insulin degludec in patients with type 2 diabetes mellitus in inadquete control on oral antidiabetic drug (OAD) therapy or OAD Therapy in combination with basal insulin.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years (both inclusive) at the time of signing informed consent form (ICF)
2. Body mass index between 18.5 and 35.0 kg/m2 (both inclusive)
3. Diagnosed with type 2 diabetes mellitus above or equal to 6 months
4. 7.5% ≤ HbA1c ≤ 10.0% at screening.

Exclusion Criteria:

1. Female who is pregnant, breast-feeding.
2. Presence or history of malignant neoplasm prior to screening.
3. Diabetic ketoacidosis, diabetic lactic acidosis, or diabetic nonketotic hyperosmolar syndrome within 6 months prior to screening.
4. Known or suspected hypersensitivity to investigational medical product(s) or related products.
5. Severe hypoglycemia (Level 3 hypoglycemia) within 6 months prior to screening
6. History of acute heart failure within 6 months prior to screening or hospitalization for coronary heart disease, myocardial infarction, unstable angina, stroke within 6 months prior to screening.
7. Participation in a clinical study of another study drug within 3 month prior to randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2024-07-13 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | From baseline (week 0) to week 16
  Change from baseline in HbA1c after 16 weeks of treatment

SECONDARY OUTCOMES:
Change in fasting plasma glucose(FPG) | From baseline (week 0) to week 16
  Change from baseline in fasting plasma glucose (FPG) after 16 weeks of treatment
Weekly doses of GZR4 Injection/Insulin Degludec | Week 15-16
  Weekly doses of once-weekly GZR4 Injection and once-daily Insulin Degludec Injection from week 15 to week 16 are presented.
Incidence and Rate of Treatment-emergent adverse events (TEAEs) | From baseline (week 0) to week 20
  A TEAE is defined as an event that had onset date (or increase in severity) during the on-treatment observation period.
Incidence and Rate of hypoglycemia episodes | From baseline (week 0) to week 20
  Hypoglycaemia alert episodes (level 1) are defined as episodes that are sufficiently low for treatment with fast-acting carbohydrate and dose adjustment of glucose-lowering therapy with plasma glucose value of equal to or above (>=) 3.0 and less than (<) 3.9 mmol/L (>= 54 and < 70 mg/dL) confirmed by blood glucose (BG) meter. Clinically significant hypoglycaemic episodes (level 2) are defined as episodes that are sufficiently low to indicate serious, clinically important hypoglycaemia with plasma glucose value of less than (<) 3.0 mmol/L (54 mg/dL). Severe hypoglycaemic episodes (level 3) are defined as episodes that were associated with severe cognitive impairment requiring external assistance for recovery. Severe hypoglycaemic episodes (level 3) are defined as episodes that are associated with severe cognitive impairment requiring external assistance for recovery.
Change in ADA of GZR4 | From baseline (week 0) to week 16
  Blood samples will be analysed for anti-GZR4 antibodies
Change in Nab of GZR4 | From baseline (week 0) to week 16
  Blood samples will be analysed for Nab

CONTACTS AND LOCATIONS:
Overall Officials: Chunyue Hao, Study Director — Gan & Lee Pharmaceuticals.
Locations (8):
- China (8):
  - Study Site 07, Wuhan, Hubei
  - Study Site 06, Changzhou, Jiangsu
  - Study Site 08, Jinan, Shandong
  - Study Site 04, Zibo, Shandong
  - Study Site 03, Xi’an, Shanxi
  - Study Site 02, Beijing
  - Study Site 05, Beijing
  - Study Site 01, Tianjin

IPD SHARING:
Plan to Share IPD: No